CLINICAL TRIAL: NCT03894644
Title: Knowledge Transfer and Retention of Simulation-based Learning for Neurosurgical Instruments: a Randomized Trial of 100 Perioperative Nurses
Brief Title: Simulation-based Learning for Neurosurgical Instruments in Perioperative Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, David Clarke, Neurosurgeon, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 100 Nurses
Record Dates: First submitted 2019-03-21; First posted 2019-03-28 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Focus of Study: Simulation Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: simulation training before instruments (Experimental): Group A performed simulation training before the recognition of real surgical instruments.
  Interventions: Other: Simulation technology
- Group B:instruments before simulation training (Active Comparator): Group B performed the recognition of real surgical instruments without prior simulation training.
  Interventions: Other: Simulation technology

INTERVENTIONS:
Other: Simulation technology — The intervention involves three consecutive sessions of the PeriopSim™ Instrument Trainer, followed by two consecutive sessions of the PeriopSim™ for Burr Hole Surgery (https://periopsim.com).

SUMMARY:
Rapid technological advances in the last 20 years have led to the exponential adoption of simulation-based learning in nursing education.

DETAILED DESCRIPTION:
Simulation-based learning is designed to engage, challenge and enrich the learner's knowledge base and skill set. It presents the opportunity to experience a variety of clinical scenarios, both common and uncommon, in a safe environment allowing repeated skills training and facilitating the transfer of classroom-knowledge to real situations.Research demonstrates that simulation can improve student engagement and learning and is being increasingly used as an educational strategy for nursing students. This prospective randomized controlled study that was undertaken with the following goals:

1. to investigate the effectiveness of simulation-based training in a large sample of perioperative nurses, measured as nurses' learning progress in the simulation environment;
2. to determine whether the learning acquired through this training is transferable to recognizing real surgical instruments; and
3. to evaluate whether simulation-based learning is retained at least one week.

ELIGIBILITY:
Inclusion Criteria:

* Perioperative nurse
* Employed at Queen Elizabeth II Health Sciences Center

Exclusion Criteria:

-Unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
Change in time saved for simulation task | Day 1 and Day 7
  Time saved is defined as the duration in seconds from the time the participant correctly submits an instrument prior to the maximum allotted time. Change is measured over repeated sessions on Day 1 and Day 7.
Change in number of errors for simulation task | Day 1 and Day 7
  Number of errors are counted as the number of incorrectly selected instruments on the first attempt. Change is measured over repeated sessions on Day 1 and Day 7.
Change in total score for simulation task | Day 1 and Day 7
  Total score is a gamification-based algorithm dependent upon the number of correct responses in the first attempt and time saved. Change is measured over repeated sessions on Day 1 and Day 7.
Difference in total score for knowledge transfer task | Day 7
  Score is defined as the number of correctly identified instruments from the instrument tray during the instrument recognition task. The difference in score is measured between arms.
Difference in time for knowledge transfer task | Day 7
  Time is the number of seconds (to a maximum of 45) taken to complete the real instrument task. The difference in score is measured between arms.

CONTACTS AND LOCATIONS:
Overall Officials: David Clarke, Principal Investigator — NSHA

IPD SHARING:
Plan to Share IPD: No